CLINICAL TRIAL: NCT06259890
Title: Sodium Intake in spondyLoarthriTes: Analysis of the Influence on the Activity of the Disease and the Therapeutic Response to Anti IL-17A Agents.
Brief Title: Influence of Sodium Intake in spondyLoarthriTes
Acronym: SALT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Collaborators: French Society of Rheumatology (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2023/807
Record Dates: First submitted 2024-01-31; First posted 2024-02-14 (Actual); Last update posted 2025-07-09 (Actual); Status verified 2024-11

CONDITIONS: Spondyloarthritis, Axial; Arthritis, Psoriatic
Keywords: Sodium intake
MeSH Terms: conditions — Axial Spondyloarthritis; Arthritis, Psoriatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Patients with radiographic/non-radiographic Axial Spondylitis or psoriatic arthritis (Other): Patients with radiographic/non-radiographic Axial Spondylitis or psoriatic arthritis managed in the rheumatology departments of the study centres.
  Interventions: Other: measurement of salt intake

INTERVENTIONS:
Other: measurement of salt intake — measurement of salt intake without intervention

SUMMARY:
The aim of the SALT study is to analyze the relationship between dietary sodium intake and disease activity in patients with axial spondyloarthritis (radiographic or non-radiographic) or psoriatic arthritis.

ELIGIBILITY:
Inclusion Criteria:

* patients with axial spondyloarthritis (radiographic or non-radiographic) or psoriatic arthritis
* women who have been menopausal for at least 24 months, surgically sterilized, or, for women of childbearing potentiale, use an effective method of contraception (oral contraceptives, contraceptive injections, intrauterine devices, double-barrier method, contraceptive patches)

Exclusion Criteria:

* patient treated by cyclosporine, diuretics, angiotensin-converting enzyme inhibitors or angiotensin II receptor antagonists.
* current treatment with an anti-IL-17A agent (secukinumab or ixekizumab or bimekizumab or brodalumab) or with an anti-IL23 agent (ustekinumab, guselkumab, risankizumab or tildrakizumab) or previous treatment less than 6 months old.
* patients on systemic corticosteroids with corticosteroid therapy > 10 mg prednisone equivalent
* pregnant woman

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2024-01-30 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
sodium intake | day of inclusion, monday and tuesday following
  average sodium concentration in urine for the week

CONTACTS AND LOCATIONS:
Locations (4):
- France (4):
  - CHU Besançon, Besançon
  - CHD Vendée, La Roche-sur-Yon
  - CHU St Etienne, Saint-Etienne
  - Hôpital Nord Franche-Comté, Trévenans

IPD SHARING:
Plan to Share IPD: No